CLINICAL TRIAL: NCT02049398
Title: Temporal Variation In The Oral Microbiome
Brief Title: Study of Variation Over Time in the Oral Microbiome
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999914047; 14-C-N047
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Microbiota; Oral Health; Body Mass Index
Keywords: Microbiome; Saliva; Reliability; Oral Cavity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Oral microbiome cohort: a cohort of 40 adults willing to provide oral samples approximately every two months forone year

SUMMARY:
Background:

- Normal bacteria and other tiny organisms are found in healthy human mouths. These are called oral microbiota. It is unclear exactly how the oral microbiota may affect health. For example, if the microbial composition is abnormal, it may lead to mouth conditions like periodontitis. Researchers want to study how the microbiota changes over time. This can help them plan future disease studies.

Objectives:

- To see if and how oral microbiota change over time.

Eligibility:

- Forty adult employees of the National Cancer Institute Shady Grove.

Design:

* For 12 hours before the first visit, participants will not eat or drink (except water). They will not brush, floss, use mouthwash, chew gum, eat lozenges or candies, smoke cigarettes, or chew tobacco.
* At the first visit, participants will:
* Be given a saliva collector. They will spit 2 mL of saliva into it.
* Fill out an online questionnaire.
* Every 2 months, participants will visit the clinic and repeat visit 1.
* The study ends after 1 year.

Sponsoring Institute: National Cancer Institute

DETAILED DESCRIPTION:
The Human Microbiome Project (HMP), started in 2008, aimed to characterize the microbial communities on the skin, in the oral and nasal cavities, and in the gastrointestinal and urogenital tracts. This project cross-sectionally described the microbial communities in a healthy human population, but did not adequately describe longitudinal stability. Out of the 236 adults included in the HMP, a second saliva sample was collected on a small subset (N=74) with a long interval between collections, an average of 203 days. Community similarity was calculated between two visits; for saliva samples, the Spearman correlation was high (rs=0.8). However, it was unclear which metric of community similarly was being used for this calculation. When we obtained the HMP data and calculated the Spearman correlation for specific diversity metrics in the saliva samples, the correlations were weaker and ranged from 0.225 to 0.524 for the Shannon Index and PD tree, respectively. Other studies with fewer people, but more time points, have had conflicting conclusions on the temporal variation of the oral microbiome. Given this variability, it is vital to establish whether a single measurement is representative of the typical composition of microbiota in a specific body site using more than two time points.

In epidemiological studies, it is often impractical, if not impossible, to collect biological samples or measurements multiple times for each participant during the study period. However, when a biological sample or a measurement is taken only once, there is concern that the single assessment is not representative of the typical value. For example, serum 25(OH)D levels, which are used to assess an individual s vitamin D exposure, have seasonal fluctuations, but studies have established that a single measurement is sufficiently reliable to represent typical exposure. The correlation between samples over time is also used to create more accurate power calculations for future studies.

Since previous work has not adequately addressed temporal variation in the oral microbiome, we propose to: 1) establish a cohort of 40 adults willing to provide oral samples approximately every two months for one year; 2) process all oral samples and evaluate the presence and quantity of microbiota using 16S ribosomal RNA gene sequencing; 3) calculate appropriate reliability measures for the sample over time using the intra-class correlation coefficient (ICC) for and <= diversity metrics; and 4) empirically evaluate the efficiency of different longitudinal designs including two or more sample collections with an outcome such as body mass index (BMI). Because of the complexity and high prevalence of human DNA in saliva, metagenomic analyses of oral samples are not yet feasible, however, the samples obtained from this study will be available for use in future metagenomic analyses when the technology is operationalized. The current study is essential to establish the reliability of a single measure of the oral microbiome to determine appropriate sample sizes for future cohort studies considering the effect of the oral microbiome on the risk of cancer and other health outcomes.

ELIGIBILITY:
* Everyone who plans to continue working at the NCI for at least a year is eligible to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Employees of the National Cancer Institute.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2014-01-28 (Actual); Primary Completion 2015-09-16 (Actual); Study Completion 2015-12-23 (Actual)

PRIMARY OUTCOMES:
Intraclass correlation coefficient for alpha/beta diversity measures. | 10 months
  Stability of oral microbiome over 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian Abnet, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Zhou Y, Gao H, Mihindukulasuriya KA, La Rosa PS, Wylie KM, Vishnivetskaya T, Podar M, Warner B, Tarr PI, Nelson DE, Fortenberry JD, Holland MJ, Burr SE, Shannon WD, Sodergren E, Weinstock GM. Biogeography of the ecosystems of the healthy human body. Genome Biol. 2013 Jan 14;14(1):R1. doi: 10.1186/gb-2013-14-1-r1. PMID 23316946
- [Background] Costello EK, Lauber CL, Hamady M, Fierer N, Gordon JI, Knight R. Bacterial community variation in human body habitats across space and time. Science. 2009 Dec 18;326(5960):1694-7. doi: 10.1126/science.1177486. Epub 2009 Nov 5. PMID 19892944
- [Background] Lazarevic V, Whiteson K, Hernandez D, Francois P, Schrenzel J. Study of inter- and intra-individual variations in the salivary microbiota. BMC Genomics. 2010 Sep 28;11:523. doi: 10.1186/1471-2164-11-523. PMID 20920195